CLINICAL TRIAL: NCT01741051
Title: A Randomized Air Filter Intervention Study of Air Pollution and Fetal Growth in a Highly Polluted Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Simon Fraser University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Ryan Allen, Associate Professor, Simon Fraser University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 275997
Record Dates: First submitted 2012-11-30; First posted 2012-12-04 (Estimated); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Fetal Growth Restriction
Keywords: Air pollution; Particulate matter; Mongolia; Pregnancy; Intrauterine growth restriction (IUGR); Fetal growth; Birth weight; Gestational age; Obesity; IQ; Autism; Wheeze
MeSH Terms: conditions — Fetal Growth Retardation; Birth Weight; Obesity; Autistic Disorder; Respiratory Sounds

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HEPA Filter (Experimental): HEPA filter(s) placed in the participant's home from approximately 10 weeks gestation until birth.
  Interventions: Device: HEPA Filter
- Control (No Intervention)

INTERVENTIONS:
Device: HEPA Filter
  Arms: HEPA Filter

SUMMARY:
The purpose of this study is to use an air filter intervention to evaluate the relationship between particulate matter air pollution exposure during pregnancy and fetal growth. We hypothesize that: 1) portable high efficiency air (HEPA) filters will produce major reductions in home indoor concentrations of particulate matter and 2) pregnant women whose exposures to particulate matter are reduced by this intervention will give birth to children with greater mean body weight for gestational age.

In an extended follow-up of this cohort, we aim to evaluate the relationship between use of portable air purifiers during pregnancy and the growth and development of children from birth to age four years. In particular, the follow-up study will focus on children's physical growth, respiratory symptoms, and behavioral, social and neurocognitive development.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 years)
* Pregnant woman in first trimester (<14 weeks)
* Single gestation pregnancy
* Non-smoker

Exclusion Criteria:

* Multiple-gestation pregnancy
* Current smoker
* Currently operating an air filter in the home
* Currently living in a ger (traditional Mongolian felt-lined yurt)
* Plan to give birth outside of a hospital or clinic in Ulaanbaatar

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 540 (Actual)
Dates: Start 2014-01; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Gestational-age adjusted birthweight | At birth
Birthweight | At birth
Gestational age | At birth
Head circumference | At birth
Small for gestational age | At birth
  <10%ile of birth weight for gestational age
Birth length | At birth
  Birth length
Child body mass index | Age 2 years
  BMI = weight(kg)/height(m)^2
Child body mass index | Age 4 years
  BMI = weight(kg)/height(m)^2
Child wheeze | Annually from birth to age 4 years
  Parent-reported wheeze (ever/never and phenotypes)
Child behavioural development | Age 2 years
  Sub-scales and composite scores from the Behavior Assessment System for Children, Third Edition (BASC-3)
Child behavioural development | Age 4 years
  Sub-scales and composite scores from the Behavior Assessment System for Children, Third Edition (BASC-3)
Child neurocognitive development | Age 4 years
  Sub-scales and index scores from the Wechsler Preschool and Primary Scale of Intelligence, Fourth Edition (WPPSI-IV)
Child social development | Age 4 years
  Social Responsiveness Scale, Second Edition (SRS-2) scores

SECONDARY OUTCOMES:
Blood pressure | At approximately 10, 11, 30 and 31 weeks gestation
C-reactive protein | At approximately 10 and 30 weeks gestation
Stratified Analyses | Various
  For all variables, we will explore effect modification by maternal exposure to environmental tobacco smoke, fraction of time spent at home, sex of the baby, season of birth, gestational age at birth, and the fraction of time that the HEPA filter(s) were used.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Allen, PhD, Principal Investigator — Simon Fraser University
Locations (1):
- Mongolia National University of Medical Sciences, Ulaanbaatar, Mongolia

REFERENCES:
- [Derived] Enkhbat U, Gombojav E, Banzrai C, Batsukh S, Boldbaatar B, Enkhtuya E, Bellinger DC, Lanphear BP, McCandless LC, Allen RW. Portable HEPA filter air cleaner use during pregnancy and children's autistic behaviors at four years of age: The UGAAR randomized controlled trial. Environ Int. 2022 Oct;168:107432. doi: 10.1016/j.envint.2022.107432. Epub 2022 Jul 25. PMID 36007302
- [Derived] Ulziikhuu B, Gombojav E, Banzrai C, Batsukh S, Enkhtuya E, Boldbaatar B, Bellinger DC, Lanphear BP, McCandless LC, Tamana SK, Allen RW. Portable HEPA Filter Air Cleaner Use during Pregnancy and Children's Cognitive Performance at Four Years of Age: The UGAAR Randomized Controlled Trial. Environ Health Perspect. 2022 Jun;130(6):67006. doi: 10.1289/EHP10302. Epub 2022 Jun 22. PMID 35730943
- [Derived] Enkhbat U, Gombojav E, Banzrai C, Batsukh S, Boldbaatar B, Enkhtuya E, Ochir C, Bellinger DC, Lanphear BP, McCandless LC, Allen RW. Portable HEPA filter air cleaner use during pregnancy and children's behavior problem scores: a secondary analysis of the UGAAR randomized controlled trial. Environ Health. 2021 Jul 5;20(1):78. doi: 10.1186/s12940-021-00763-6. PMID 34225757
- [Derived] Barn P, Gombojav E, Ochir C, Boldbaatar B, Beejin B, Naidan G, Galsuren J, Legtseg B, Byambaa T, Hutcheon JA, Janes C, Janssen PA, Lanphear BP, McCandless LC, Takaro TK, Venners SA, Webster GM, Allen RW. The effect of portable HEPA filter air cleaner use during pregnancy on fetal growth: The UGAAR randomized controlled trial. Environ Int. 2018 Dec;121(Pt 1):981-989. doi: 10.1016/j.envint.2018.08.036. Epub 2018 Sep 10. PMID 30213473